CLINICAL TRIAL: NCT03353779
Title: The Impact Of Platelet Function on 1-year Outcome in Complex PCI Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Yi-Da Tang, Professor, Chief Physician, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 2017-901
Record Dates: First submitted 2017-11-20; First posted 2017-11-27 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Percutaneous Coronary Intervention; Coronary Artery Disease
Keywords: Percutaneous coronary intervention; antiplatelet; platelet function; prognosis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To identify the optimal cut-off values in different platelet function testing to predict MACCE at 12-months in complex PCI patients of China

DETAILED DESCRIPTION:
This study will observe the relationship between platelet function testing and clinical outcomes. Meanwhile we aim to identify optimal cut-off values in different platelet function testing, including IPF, TEG and VerifyNow, to predict MACCE during12-months in complex PCI patients.

ELIGIBILITY:
Inclusion Criteria:

* Documented undergoing complex PCI in 1 year prior to enrollment.

Exclusion Criteria:

* Presence of any condition/circumstance which in the opinion of the investigator could significantly limit the complete follow up of the patient (e.g. tourist, non-native speaker or does not understand the local language where interpreter services are not reliably available, psychiatric disturbances, alcohol or drug abuse).
* Presence of serious/severe co-morbidities in the opinion of the investigator which may limit life expectancy (<1 year).
* Current participation in a blinded randomized clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with complex PCI were defined as having at least 1of the following features :3 vessels treated,≥3 stents implanted, ≥3 lesions treated,bifurcation with 2stents implanted ,total stent length >60 mm or chronic total occlusion.
Sampling Method: Non-Probability Sample
Enrollment: 1440 (Estimated)
Dates: Start 2017-11-29 (Actual); Primary Completion 2021-07-29 (Estimated); Study Completion 2021-07-29 (Estimated)

PRIMARY OUTCOMES:
Optimal cut-off values in different platelet function testing to predict MACCE at 12-months in complex PCI patients of China | Within 12 months of patient enrolled

SECONDARY OUTCOMES:
Effectiveness and sensitivity of predicting between different platelet function testing | Within 12 months of patient enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Yida Tang, MD, PhD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Chinese Academy of Medical Sciences Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided